CLINICAL TRIAL: NCT07076381
Title: New at Parenting Study
Acronym: NAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of San Francisco (Other)
Responsible Party: Principal Investigator, Dhara Meghani, Associate Professor, University of San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 934
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Control Group; Counseling
Keywords: Teletherapy; Brief therapy; Postpartum Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control group participants will have an assigned counselor for the study duration and can access them at any time. They will not have a defined treatment schedule in the way that counseling group participants do.
- Counseling Group (Experimental): Counseling group participants will receive three brief therapy sessions virtually from the same counselor between 1 and 5 months postpartum. The intervention is adapted from brief and solutions-therapy and operates on single-session therapy principles.
  Interventions: Behavioral: Brief and solutions-therapy intervention

INTERVENTIONS:
Behavioral: Brief and solutions-therapy intervention — Parents will receive three phone counseling sessions over "Zoom" of 45-60 minutes each from a counselor when their baby is 4-6 weeks old; 10-12 weeks old, and 16-20 weeks old. The date and time of the sessions will be coordinated by phone or e-mail between the parent and their counselor in the week preceding the call. Following their session, parents in this group will receive a brief satisfaction survey over e-mail (Appendix E) that they will be asked to complete within 72 hours.
  Arms: Counseling Group

SUMMARY:
This study examines whether a brief counseling intervention provided to parents virtually in the first six months after having their baby is able to reduce and prevent the development of depression symptoms, anxiety, and stress. It also explores whether parents' confidence increases over time and whether they feel more support by the end of the intervention. The study will compare a group of parents who receive the intervention from trained graduate students in clinical psychology with a group of parents who do not receive the intervention.

Select parents will also be interviewed to understand their experiences of new parenting and to help explain the research findings of the study.

DETAILED DESCRIPTION:
The primary purpose of this pilot study is to examine the impact of receiving regularly scheduled phone counseling services delivered by advanced, trained clinical psychology doctoral students during the first six months of parenthood, for low-risk first-time parents. This study will examine whether parents who receive scheduled phone counseling services delivered through brief therapy techniques demonstrate a greater change from pregnancy to six months postpartum in their anxiety symptoms, depressive symptoms, self-efficacy/parenting confidence, stress, and social support when compared to a matched control group of parents who do not receive regularly scheduled phone calls.

A secondary purpose of this study is to qualitatively explore the experience of parents who undergo the initial transition to parenthood; that is, what are the common themes requiring support that emerge with respect to the transition to parenthood? Additionally, the study aims to identify the acceptability and utility of using a phone-based counseling service for new parents and to elicit feedback about potential modifications that can be made to increase the positive impact of the service in the future.

ELIGIBILITY:
Inclusion Criteria:

* Biological parent who is (or has a partner who is) between 27 and 39 weeks pregnant with first child OR a parent who is planning to adopt a newborn child within the timeline of the study;
* Parent does not have current psychiatric history/hospitalizations;
* Parent has a reliable phone and/or computer connection that will enable them to receive calls from Parentline team member and complete online questionnaires

Exclusion Criteria:

Participants who do not meet the inclusion criteria will not be eligible for the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Postpartum Specific Anxiety Scale | At 1 month and 6 months postpartum
  This 51-item self-report scale is designed to examine the frequency, and not severity, of anxieties specific to the postpartum period. The PSAS is not a diagnostic tool, nor is it to be used for screening purposes, at present. The PSAS was developed and validated for use with mothers of infants aged between 0 and 6 months. The PSAS includes items about emotional distress, and anxieties related to the participant's newborn infant.
Edinburgh Postnatal Depression Scale | At enrollment, 1 month postpartum, and 6 months postpartum
  The EPDS assesses depressive symptoms in the past week using a 4-point likert scale. Total scores range from 0 to 30 and a cutoff score of 10 or 13 is commonly used to indicate possible depression.
Perceived Stress Scale - Short Form | At enrollment, 1 month postpartum, and 6 months postpartum
  The PSS is a 10-item measure commonly used to measure the degree of "how unpredictable, uncontrollable, and overloaded respondents find their lives."
Karitane Parenting Confidence Scale | At 1 month postpartum and 6 months postpartum
  The scale measures self-efficacy among parents of infants 0 through 12 months of age. Respondents answer 15 items on a 4-point likert scale; a score of 39 or less is indicative of low levels of parenting confidence.
Multidimensional Scale of Perceived Social Support | At enrollment, 1 month postpartum, and 6 months postpartum
  The Multidimensional Scale of Perceived Social Support is a measure of how much support a parent feels they get from family, friends and significant others.
State-Trait Anxiety Inventory - Short Form | At enrollment
  This is a 6-item measure of how participants are feeling in the moment.

SECONDARY OUTCOMES:
Brief Infant Sleep Questionnaire | At 6 months postpartum
  This is a screening tool that can be used to identify sleep concerns in infants.

CONTACTS AND LOCATIONS:
Overall Officials: Dhara Meghani, PhD, Principal Investigator — University of San Francisco
Locations (1):
- University of San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
This is a pilot study with a small data set. We will make it available for public use or by request on a public data repository.
Time Frame: Start date: July 15, 2025 End date: N/A
Access Criteria: Other researchers will be able to access a de-identified data set with three time points of data from both groups in the study. They will also have access to the primary outcome measures used in order to see how the data were scored. They can access these materials on Open Science Framework
URL: https://doi.org/10.17605/OSF.IO/7STHM

REFERENCES:
- See also: Related Info — https://doi.org/10.17605/OSF.IO/7STHM
- Available data/document: Individual Participant Data Set: https://doi.org/10.17605/OSF.I — https://osf.io/dashboard — Open Science Framework website for Principal Investigator, which includes public access to de-identified data set